CLINICAL TRIAL: NCT04559919
Title: Prospective Regional Epilepsy Database and Biobank for Individualized Clinical Treatment
Brief Title: Prospective Regional Epilepsy Database
Acronym: PREDICT
Status: Recruiting | Type: Observational
Sponsor: Sahlgrenska University Hospital (Other)
Responsible Party: Principal Investigator, Johan Zelano, Consultant Neurologist, Sahlgrenska University Hospital
Other Study IDs: 2020-00853
Record Dates: First submitted 2020-09-08; First posted 2020-09-23 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Epilepsy
Keywords: epilepsy; biomarker; access to care; quality of care; seizure
MeSH Terms: conditions — Epilepsy; Seizures | interventions — Demography; Delivery of Health Care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Biospecimen Retention: Samples With DNA — Blood samples, and for some individuals cerebrospinal fluid (if lumbar puncture is indicated for clinical reasons, extra csf will be collected).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Adults with epilepsy: Adults over 18 years of age, with an unprovoked seizure in the last year or epilepsy, resident in VGR at the time of inclusion. Languages available: Swedish, English, Arabic.
  Based on the clinical information, patients can be categorized into relevant groups; single seizure, seizure-free with epilepsy, and drug-resistant epilepsy. Subgroups may also be selected based on age, sex, epilepsy sub-diagnosis, cause of epilepsy, use of a particular antiepileptic drug, or experience of a particular side effect.
  Interventions: Other: Seizure status; Diagnostic Test: Tests; Other: Epilepsy; Other: Demographics and psychosocial; Other: Health care

INTERVENTIONS:
Other: Seizure status — We will collect information on first seizure ever, last seizure ever, number of seizure in last two months.
Diagnostic Test: Tests — We will collect results from imaging, electroencephalogram, and laboratory tests.
Other: Epilepsy — We will collect information on risk factors of epilepsy, cause of epilepsy, epilepsy type/syndrome, medications tried, if the epilepsy is drug resistent, side effects of antiepileptic drugs.
Other: Demographics and psychosocial — We will collect information on age, sex, date of death if applicable, marital status, education level, income type, driving status, employment, benefits, sick leave, number of household members.
Other: Health care — We will collect information on received health care; visit dates, caregiver, dispensation dates of antiepileptic drugs

SUMMARY:
PREDICT is an observational study following adults with an unprovoked seizure or epilepsy in the health care region of western Sweden. The objective is to identify biomarkers and/or genetic predisposition of relevance for diagnosis and/or treatment of epilepsy and study the long-term prognosis and consequences of epilepsy.

DETAILED DESCRIPTION:
Adults over 18 years of age, with an unprovoked seizure in the last year or epilepsy, resident in the health care region of western Sweden (VGR) at the time of inclusion.

Baseline data and outcome variables are collected from several patient registries: the electronic medical records system in the health care region VGR and Swedish National Registers of healthcare, income, and employment managed by The National Board of Health and Welfare or Statistics Sweden, both of which are government agencies.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years of age
* An unprovoked seizure within the last year or a diagnosis of epilepsy according to the current International League Against Epilepsy definition (epilepsy with seizure in the last ten or antiepileptic drug treatment in the last five years)

Exclusion Criteria:

* Expected survival less than two years
* Inability to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with an unprovoked seizure or epilepsy, resident in VGR at inclusion.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2020-11-27 (Actual); Primary Completion 2031-12-31 (Estimated); Study Completion 2031-12-31 (Estimated)

PRIMARY OUTCOMES:
epilepsy | baseline and years 1,2,3,4,5,6,7,8,9,10
  more than one seizure after first seizure
seizure status | baseline and years 1,2,3,4,5,6,7,8,9,10
  the number of seizures in last two months and overall
drug resistant epilepsy | baseline and years 1,2,3,4,5,6,7,8,9,10
  epilepsy that has not responded to two antiepileptic drugs
severe side effects of antiepileptic drug | baseline and years 1,2,3,4,5,6,7,8,9,10
psychosocial outcomes | baseline and years 1,2,3,4,5,6,7,8,9,10
  employment, marital status, income, sick leave

SECONDARY OUTCOMES:
received health care | baseline and years 1,2,3,4,5,6,7,8,9,10
  the number of visits for epilepsy, missed appointments, time intervals between visits

CONTACTS AND LOCATIONS:
Overall Officials: Johan Zelano, MD PhD, Principal Investigator — Sahlgrenska University Hospital
Locations (3):
- Sweden (3):
  - Södra Älvsborgs Sjukhus, Borås
  - Sahlgrenska University Hospital, Gothenburg
  - Sjukhusen i Väster, Gothenburg

IPD SHARING:
Plan to Share IPD: No
The data will be protected by privacy laws and cannot be shared even if anonymized, because of the high resolution of data.

REFERENCES:
- [Derived] Andersson K, Akel S, Asztely F, Larsson D, Zetterberg H, Zelano J. Higher plasma total tau concentrations among patients reporting CNS-related side effects from antiseizure medication. Seizure. 2025 Feb;125:99-105. doi: 10.1016/j.seizure.2025.01.015. Epub 2025 Jan 13. PMID 39826304